CLINICAL TRIAL: NCT04547673
Title: To Develop and Validate a Nasoendoscopic Intelligent Diagnostic System for Nasopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weiping Wen, Vice President of First Affiliated Hospital, Sun Yat-Sen University; President of sixth Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZSYY2020
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Otolaryngological Disease; Artificial Intelligence
Keywords: Nasopharyngeal Carcinoma; Endoscopy; Narrow-Band Imaging; White-Light Imaging
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NPC group: Patients pathologically diagnosed as NPC by agreement of 2 experienced pathologists who were blinded to the corresponding endoscopic assessment.
  Interventions: Diagnostic Test: rigid nasal endoscopes
- Non-NPC group: Patients pathologically diagnosed as non-NPC (including inflammatory hyperplasia, Atypical hyperplasia, Papilloma etc.) by agreement of 2 experienced pathologists who were blinded to the corresponding endoscopic assessment.
  Interventions: Diagnostic Test: rigid nasal endoscopes

INTERVENTIONS:
Diagnostic Test: rigid nasal endoscopes — The endoscope is introduced through the nasal passage to observe, in sequence, the posterior nostril, superior and posterior walls of the nasopharynx, torus tubarius, pharyngeal opening of the auditory tube, and Rosenmu¨ller recess. The imaging light mode is set to conventional WLI and subsequently switch to NBI during the procedure, and representative images are collected and preserve for further analysis. All lesions, detected by either WLI or NBI, are biopsied.

SUMMARY:
Nasopharyngeal carcinoma (NPC) occurs at a high frequency in southern China, northern Africa, and Alaska, with a reported incidence of 30 cases per 100 000 in Guangdong Province. Endoscopic examination and biopsy are the main methods used for detection and diagnosis of NPC. Early NPC patients achieve favourable prognoses after concurrent radiotherapy and chemotherapy in compassion with advanced NPC patients.

Here, the investigators focused on the utility of artificial intelligence to detect early NPC, which based on white light imaging (WLI) and Narrow-band imaging (NBI) nasoendoscopic examination. Having access to this unique population provides an unprecedented opportunity to investigate the effect of intelligent system on diverse nasopharyngeal lesions detection and develop a novel Computer-Aided Diagnosis System.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age

Exclusion Criteria:

* Refuse to sign the informed consent statement
* Patients who have contraindications, e.g. coagulation dysfunction, drug allergy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at the outpatient department of otolaryngology at the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, People's Republic of China, or patients at Sun Yat-Sen University Cancer Center and Kiang Wu Hospital, with risk factors including any of the following: Cantonese ethnicity, NPC family history, Epstein-Barr virus detection, any symptom of nasal obstruction, sense of peculiar smell, blood-stained nasal discharge, epistaxis, ear fullness, tinnitus, hearing loss, diplopia, headache, or cervical mass.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological diagnosis | baseline
  All lesions, detected by either WLI or NBI, are biopsied. 2 experienced pathologists, who were blinded to the endoscopic and intelligent assessment, evaluate the pathological nature of the biopsied lesion independently, and 2 professors with over 10 years of experience in Otolaryngology and pathology department are consulted in cases of disagreement.

SECONDARY OUTCOMES:
Lesion range | baseline
  All images in which lesions are pathologically diagnosed as NPC are collected. 2 experienced pathologists, who were blinded to the endoscopic and intelligent assessment, delineated the malignant area in the images independently, and 2 professors with over 10 years of experience in Otolaryngology department are consulted in cases of disagreement.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Wen, Ph.D, Study Director — Otolaryngology Department, First Affiliated Hospital of Sun Yat-sen University
Locations (3):
- China (3):
  - First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Kiang Wu Hospital, Macao, Macao

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He R, Jie P, Hou W, Long Y, Zhou G, Wu S, Liu W, Lei W, Wen W, Wen Y. Real-time artificial intelligence-assisted detection and segmentation of nasopharyngeal carcinoma using multimodal endoscopic data: a multi-center, prospective study. EClinicalMedicine. 2025 Feb 15;81:103120. doi: 10.1016/j.eclinm.2025.103120. eCollection 2025 Mar. PMID 40026832